CLINICAL TRIAL: NCT03203031
Title: Postoperative Pain in Neonates After Abdominal Surgery Using Ultrasound Guided Quadratus Lumborum Block Performed at the Beginning of the Procedure
Brief Title: Postoperative Pain in Neonates After Abdominal Surgery Using Quadratus Lumborum Block
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hôpital Armand Trousseau (Other)
Responsible Party: Principal Investigator, Pr Isabelle CONSTANT, Professor, Hôpital Armand Trousseau
Other Study IDs: CARRE DES LOMBES
Record Dates: First submitted 2017-06-19; First posted 2017-06-29 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
Keywords: pain; neonate; regional anesthesia; postoperative
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates with abdominal surgery and quadratus lumborum block: 0-6 months children with abdominal surgery. After standard induction of general anesthesia, patients will receive 0.5 ml/kg of ropivacaine (2 mg/ml) in a quadratus lumborum block. Ultrasonography will be used to guide the injection. In the postoperative period, pain scores and analgesics consumption will be recorded until the 48th hour post surgery.
  Interventions: Procedure: General anesthesia; Procedure: Quadratus lumborum block

INTERVENTIONS:
Procedure: General anesthesia — Standard general anesthesia
Procedure: Quadratus lumborum block — Guided by ultrasonography, injection of 0.5 ml/kg of ropivacaine (2 mg/ml) between the quadratus lumborum muscle and the internal oblique muscle, before skin incision

SUMMARY:
Postoperative pain scores and analgesic requirements will be evaluated in neonates after abdominal surgery, with regional quadratus lumborum block performed at the beginning of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* abdominal surgery under general anesthesia
* spontaneously breathing before the procedure

Exclusion Criteria:

* multiple organ failure
* mechanical ventilation before the procedure

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with planned abdominal surgery under general anesthesia, recruited in our neonatology unit.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | At the 24th hour after surgery
  standard pain scale used in neonatology in our institution: EDIN (Echelle Douleur Inconfort Nourrisson)
morphine consumption | At the 24th hour after surgery
  cumulative morphine dose administered to the patient
nalbuphine consumption | At the 24th hour after surgery
  cumulative nalbuphine dose administered to the patient
postoperative pain score | At the 24th hour after surgery
  standard pain scale used in neonatology in our institution: EVENDOL (EValuation ENfant Douleur)

SECONDARY OUTCOMES:
morphine consumption | At the 48th hour after surgery
  cumulative morphine dose administered to the patient
nalbuphine consumption | At the 48th hour after surgery
  cumulative nalbuphine dose administered to the patient

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Constant, MD-PHD, Study Director — Hopital Armand Trousseau, Université Paris 6, Département d'anesthésie
Locations (1):
- Hopital Armand Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided